CLINICAL TRIAL: NCT05406752
Title: An Open-label, Single Treatment, Single Period, Single Buccal Dose Pharmacokinetic Study of Paracetamol Uniflash (125 mg/ 1.25 mL) in Healthy, Adult, Human Subjects Under Fasting Conditions.
Brief Title: Pharmacokinetic Study of Paracetamol UNIFLASH (125 MG/1.25 ML)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Unither Pharmaceuticals, France (Industry)
Collaborators: Raptim Research (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UP-CLI-2021-002
Record Dates: First submitted 2022-06-01; First posted 2022-06-06 (Actual); Results first posted 2024-12-13 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-10

CONDITIONS: Acute Pain
MeSH Terms: conditions — Acute Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- paracetamol Uniflash (125 mg/ 1.25 mL) (Experimental): 1 sachet of paracetamol Uniflash 125mg / 1.25 mL
  Interventions: Drug: paracetamol Uniflash (125 mg/ 1.25 mL)

INTERVENTIONS:
Drug: paracetamol Uniflash (125 mg/ 1.25 mL) — Oromucosal solution (125 mg/ 1.25 mL) for buccal route

SUMMARY:
This study aims to assess the pharmacokinetic profile of a new paracetamol formulation (paracetamol Uniflash 125mg/1.25mL) for buccal use after single dose.

ELIGIBILITY:
Inclusion Criteria:

* Male and non-pregnant female human subjects, age 18 - 45 years.
* Body Mass Index between 18.5-30 Kg / m2 .
* Subjects with normal findings .
* Willingness to follow the protocol requirements

Exclusion Criteria:

* History of allergy or hypersensitivity intolerance to paracetamol and ethanol
* Significant history or current evidence of malignancy or chronic - infectious, cardiovascular, renal, hepatic, ophthalmic, pulmonary, neurological, metabolic (endocrine), hematological, gastrointestinal, dermatological, immunological or psychiatric diseases, or organ dysfunction;
* Lactating or nursing female subjects;
* History of difficulty in accessibility of veins in arms.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2022-07-22 (Actual); Primary Completion 2022-07-23 (Actual); Study Completion 2022-07-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Raptim Research Pvt. Ltd., Navi Mumbai, India

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Paracetamol Uniflash (125 mg/ 1.25 mL)
Started | 32
Completed | 32
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Paracetamol Uniflash (125 mg/ 1.25 mL)
Number analyzed (Participants) | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.97 (6.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 32
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  India | 32

OUTCOME MEASURES:

1. Primary Outcome: Paracetamol Peak Plasma Concentration (Cmax) After Single Dose
Description: Peak Plasma Concentration (Cmax) of paracetamol after single dose at different timepoints :
  Within 60 min before drug administration), at 1 min, 5 min, 10 min, 15 min, 20 min, 40 min, 1h, 2h, 4h, 6h, 8h, 10h and 12h post-dose
Time Frame: Up to 12 hours post dose
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Paracetamol Uniflash (125 mg/ 1.25 mL)
Number analyzed (Participants) | 32
ng/mL | 2181.04 (1148.85)

2. Primary Outcome: Paracetamol Area Under the Plasma Concentration Versus Time Curve (AUC) After Single Dose
Description: Area under the plasma concentration versus time curve (AUC) of paracetamol after single dose at different timepoints :Within 60 min before drug administration), at 1 min, 5 min, 10 min, 15 min, 20 min, 40 min, 1h, 2h, 4h, 6h, 8h, 10h and 12h post-dose
Time Frame: Up to 12 hours post dose
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | Paracetamol Uniflash (125 mg/ 1.25 mL)
Number analyzed (Participants) | 32
hr*ng/mL | 7097.07 (1378.45)

3. Secondary Outcome: Number of Treatment-related Adverse Events
Description: Occurrence and severity of adverse events (serious and non-serious adverse events)
Time Frame: Up to 12 hours
Measure: Number; unit: adverse events
Arm/Group | Paracetamol Uniflash (125 mg/ 1.25 mL)
Number analyzed (Participants) | 32
adverse events | 0

ADVERSE EVENTS:
Time Frame: 2 days
Arm/Group | Paracetamol Uniflash (125 mg/ 1.25 mL)
All-Cause Mortality (participants affected / at risk) | 0/32
Serious Adverse Events (participants affected / at risk) | 0/32
Other Adverse Events (participants affected / at risk) | 3/32
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Paracetamol Uniflash (125 mg/ 1.25 mL) (N=32)
Alanine aminotransferase increased (Hepatobiliary disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI shall not make any publication or communication, written or oral, in connection with the Study and the results of the Study, whether partial or final, without the prior written consent of the sponsor (UNITHER PHARMACEUTICALS) during, and following termination or expiration of this Clinical Study Services Agreement.

DOCUMENTS (1):
  • Study Protocol (2022-03-01): https://cdn.clinicaltrials.gov/large-docs/52/NCT05406752/Prot_000.pdf